CLINICAL TRIAL: NCT06344312
Title: Effectiveness of Yangxue Qingnao Granules in Preventing Post Thrombolytic Hemorrhage Transformation in Patients With Acute Cerebral Infarction: a Randomized Controlled Study
Brief Title: Effectiveness of Yangxue Qingnao Granules in Preventing Post Thrombolytic Hemorrhage Transformation in Patients With Acute Cerebral Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M2023551
Record Dates: First submitted 2024-03-25; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-01

CONDITIONS: Stroke, Acute Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Randomly take 2 bags of Yangxue Qingnao Granules orally during intravenous thrombolysis with ateplase, and then take 1 bag of Yangxue Qingnao Granules three times a day for a total of 2 weeks
  Interventions: Drug: Yangxue Qingnao Granules
- Control Group (Placebo Comparator): When receiving intravenous thrombolysis with ateplase, two bags of Yangxue Qingnao Granule Simulator were randomly taken orally. Afterwards, one bag of Yangxue Qingnao Granule Simulator was taken three times a day for a total of two weeks.
  Interventions: Drug: Yangxue Qingnao Granules

INTERVENTIONS:
Drug: Yangxue Qingnao Granules — When receiving intravenous thrombolysis with ateplase, two bags of Yangxue Qingnao Granule Simulator were randomly taken orally. Afterwards, one bag of Yangxue Qingnao Granule/ Simulator was taken three times a day for a total of two weeks.

SUMMARY:
Evaluate the effectiveness of Yangxue Qingnao Granules in preventing post thrombolytic hemorrhage transformation in patients with acute cerebral infarction, and explore its possible mechanism

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years old, regardless of gender
* After the onset of this disease, the National Institutes of Research Stroke Scale score was 2 ≤ NIHSS ≤ 20 points
* Patients who have developed symptoms within 4.5 hours and can receive rt PA intravenous thrombolysis treatment
* According to the 2019 Diagnosis Points for Major Cerebrovascular Diseases in China, patients with ischemic stroke were diagnosed as having a good recovery from the first or last onset (mRS score ≤ 1 point before this onset)
* Obtain the patient or their legal representative to voluntarily sign an informed consent form approved by the ethics committee.

Exclusion Criteria:

* Intracranial hemorrhagic diseases seen on cranial imaging: hemorrhagic stroke, epidural hematoma, intracranial hematoma, ventricular hemorrhage, subarachnoid hemorrhage, etc; If it is only oozing blood, the researcher can determine whether it is suitable for enrollment
* Severe consciousness disorder: NIHSS scored>1 point in the 1a consciousness level item
* After controlling the patient's blood pressure, the systolic blood pressure remains ≥ 180mmHg or the diastolic blood pressure remains ≥ 100mmHg
* Blood glucose<2.8mmol/L (random blood glucose measurement device can be used)
* Patients with severe mental disorders and dementia
* Diagnosed with severe active liver diseases, such as acute hepatitis, chronic active hepatitis, cirrhosis, etc; Or ALT or AST>2.0 x ULN
* Diagnosed with severe active kidney disease and renal insufficiency; Or serum creatinine>1.5 × ULN
* Concurrent malignant tumors or ongoing anti-tumor treatment; For subjects diagnosed with malignant tumors after enrollment, the decision to continue participating in the study can be based on the researcher's judgment and the subject's willingness
* Suffering from severe systemic diseases, with an estimated survival time of<90 days
* History of major surgery within 4 weeks prior to enrollment
* Participated in other clinical studies within the first 30 days of randomization, or is currently participating in other clinical studies
* The researcher believes that it is not suitable to participate in this clinical study
* Patients who are allergic to any ingredient in the study drug

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with mRS score ≤ 1 on the 90th day of treatment | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided